CLINICAL TRIAL: NCT03209752
Title: Prediction of 3D Effect of Brace in Adolescent and Children Idiopathic Scoliosis Treatment Using EOS Imaging System and "Anatomic Transfer".
Brief Title: Prediction of 3D Effect of Brace in Idiopathic Scoliosis Treatment Using EOS Imaging System and "Anatomic Transfer".
Acronym: EOSTransfert
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Demeure Orthopédie (Unknown); Anatoscope (Unknown); Clinical Investigation Centre for Innovative Technology Network (Network)
Responsible Party: Sponsor
Other Study IDs: DCIC15-01
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Idiopathic Scoliosis
Keywords: 3D analysis; Brace; EOS imagind system; Anatomical transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the accuracy of a new numerical method is evaluated for predicting the 3D effect of brace on idiopathic scoliosis. This method results from the combination of several innovative technologies: the EOS imaging system and the anatomical transfer developed by Anatoscope. This is an essential step in validating a digital tool that can be used in routine clinical practice.

DETAILED DESCRIPTION:
The whole process of brace production remains unchanged. In this study, the simulation software will not be used to influence the medical decision or the manufacture of the brace. In parallel with conventional production, anatomical transfer will be used in the deformed digital model of the trunk to simulate the effect of conventional brace on the spine. This modeling will be used to compare the correction of the conventional brace observed on the spine with EOS imaging system, with that simulated by the software.

EOS Tranfert study is a observationnal, prospective, monocentric, unrandomized and controlled study. This research doesn't modify care of the patient

ELIGIBILITY:
Inclusion Criteria:

* patients aged 9 to 15 years;
* with idiopathic scoliosis (left lumbar and / or right chest);
* with moderate scoliosis: Cobb angle evaluated between 15 ° and 35 °;
* requiring brace placement or renewal;
* having signed a non-objection form
* affiliated with, or receiving, social security

Exclusion Criteria:

* patient/parents who refuse to sign a non-objectiont form
* with unstable medical condition
* person deprived of liberty by judicial or administrative decision
* person under legal protection or unable to express their consent
* person hospitalized for psychiatric care

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children or adolescent idiopathic scoliosis patient
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the accuracy of the brace effect by the new anatomical transfer method in the frontal plane. | 12 month
  Difference measurement in degrees between the digital Cobb angle after simulation and the actual Cobb angle under brace after EOS radiography.

SECONDARY OUTCOMES:
Evaluation of the accuracy of the brace effect by the new anatomical transfer method on the spinal axial rotation. | 12 month
  Difference measurement in degrees between apical axial vertebral rotation angle (AVR) after simulation and the actual AVR under brace after EOS radiography.
Evaluation of the accuracy of brace effect by the new anatomical transfer method on the torsion index. | 12 month
  Difference measurement in degrees between the numerical torsion index after simulation and the actual torsion index under brace after EOS radiography.
Evaluation of the accuracy of the brace effect by the new anatomical transfer method in the sagittal plane | 12 month
  Difference measurement in degrees between kyphosis angle, digital lordosis after simulation and kyphosis angle, real lordosis under brace after EOS radiography.
Evaluation of the accuracy of ribs position of the patient under 3D digital model of brace with respect to the actual position under brace | 12 month
  Point-to-point distance between the average rib line after simulation and under brace after EOS radiography

CONTACTS AND LOCATIONS:
Overall Officials: Courvoisier Aurélien, MD, PhD, Principal Investigator — Pediatric Orthopedic department, University GrenobleHospital
Locations (1):
- Pediatric Orthopedic Department, University Hospital, Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical Investigation Centre for Innovative Technology Network website — http://www.cic-it.fr/cic-it-grenoble.php